CLINICAL TRIAL: NCT06311136
Title: Effectiveness of an Ecological Momentary Emotion Regulation Intervention Among Individuals With and Without Depressive Disorders: A Randomized-Controlled Trial
Brief Title: Effectiveness of an Ecological Momentary Emotion Regulation Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Ilka Mueller, Principal Investigator, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PEAK
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Depressive Disorder, Major; Persistent Depressive Disorder; Healthy
Keywords: Emotion Beliefs; Emotional Regulation; Positive Emotions; Affective Symptoms; Ecological Momentary Assessment; Internet-Based Intervention; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Emotional Regulation; Affective Symptoms; Depression

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial with an Intervention Group and a Control Group without an intervention.
Who Masked: Participant, Outcomes Assessor
Masking Description: During the treatment phase, both the intervention and monitoring-only control groups use a diary called "Positive Everyday Affect Knowledge". Participants are informed that the diary entries may include instructions for implementing specific emotion regulation strategies in their daily activities. However, this component of the procedure is not characterized explicitly as an intervention. This methodological consideration ensures that differences observed between the groups can be attributed to the intervention itself, rather than to differences in participants' expectations.
  Clinical interviews will be conducted blindly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants complete a valence-specific ecological momentary intervention twice daily over 14 consecutive days.
  The ecological momentary intervention is presented as the "Positive Everyday Affect Knowledge" (PEAK) diary and includes valence-specific emotion regulation strategy instructions. Participants receive reminders to complete surveys on their strongest emotions since the last assessment. Depending on the valence of this emotion, they receive instructions on how to use the strategy savoring (for positive emotions) or reappraisal (for negative emotions).
  Interventions: Behavioral: Valence-Specific Ecological Momentary Intervention
- Monitoring-only control group (No Intervention): Participants complete a valence-specific ecological momentary assessment twice daily over 14 consecutive days.
  The ecological momentary assessment is presented as the "Positive Everyday Affect Knowledge" (PEAK) diary, and only involves monitoring participants' emotional experiences and regulation. Participants receive reminders to complete surveys on their strongest emotions since the last assessment. Depending on the valence of this emotion (positive versus negative), they are asked about their emotion regulation strategies.

INTERVENTIONS:
Behavioral: Valence-Specific Ecological Momentary Intervention — The ecological momentary intervention is designed to enhance participants ability to select and effectively implement emotion regulation strategies fitting to the valence of their current emotions. Specifically, the intervention instructs participants to use the strategy of savoring to amplify their positive emotions, fostering an appreciation for the present moment. Conversely, for the attenuation of negative emotions, the intervention advocates to use the strategy of reappraisal, encouraging participants to reinterpret adverse situations in a more positive or neutral way, thus reducing their emotional impact. This targeted approach ensures that the emotion regulation strategies are not only effective but also contextually appropriate.
  Arms: Intervention group

SUMMARY:
This two-armed randomized controlled trial aims to investigate the effectiveness of an emotion regulation intervention in individuals with and without depressive disorders. The study encompasses participants diagnosed with mild to moderate major depression or persistent depressive disorder and healthy controls without a current depressive disorder.

Participants will be randomly assigned to either the intervention group, receiving a valence-specific emotion regulation intervention in daily life, or a monitoring-only control group. The valence-specific intervention supports the implementation of different emotion regulation strategies based on whether a person is experiencing mainly positive or negative emotions. In contrast, participants in the control group will solely monitor their positive and negative emotions and the strategies used to regulate them.

Outcome measures include emotion regulation ability, self-efficacy, and strategy use, depressive symptoms, positive and negative affect, and emotion beliefs (controllability, usefulness).

A second aim of the study is to compare beliefs about positive emotions and strategies to regulate them between individuals with and without current depressive disorders. Furthermore, the investigators aim to examine why individuals might choose unfavorable emotion regulation strategies even when feeling good. Therefore, another research question is, how emotion beliefs might explain emotion regulation strategy choice.

DETAILED DESCRIPTION:
Background:

Affective disorders, such as depression, have been consistently associated with deficiencies not only in the regulation of negative emotions but also in the maintenance and upregulation of positive emotions. However, the mechanisms underlying emotion regulation deficits in depressive disorders remain inadequately understood. Recently, there has been a growing interest in the role of beliefs about emotions as factors contributing to emotion regulation deficits in psychopathology. In light of this, this study seeks to explore potential differences in beliefs about positive (and negative) emotions between individuals with and without current depressive disorders. Another aim of this study is to examine how these individual differences in emotion beliefs predict the selection of emotion regulation strategies in daily life, particularly in the context of positive emotions.

Given the pivotal role that deficits in emotion regulation play in the onset and persistence of depressive disorders, this study aims to investigate whether an ecological momentary intervention, addressing both positive and negative emotion regulation, can effectively improve emotion regulation processes. Recent research suggests that distinct emotion regulation strategies may be effective for positive versus negative emotion regulation. Consequently, this study aims to evaluate the effectiveness of a smartphone-based, valence-specific emotion regulation intervention in individuals with and without current depressive disorders.

Method:

This study will enlist participants aged between 18 and 65, diagnosed with mild to moderate major depression or persistent depressive disorder, as well as healthy controls without a current depressive disorder. Individuals presenting with a current severe substance use disorder, acute suicidality, an ongoing severe major depressive episode, a history of bipolar disorder, or lifetime psychotic disorders are precluded from participation in both groups. Additional exclusion criteria for participation within the control cohort encompass (a) occurrence of a major depressive episode in the preceding 12 months, (b) history of severe major depressive episodes, (c) diagnosis of recurrent depressive disorder or history of persistent depressive disorder, and (d) ongoing treatment modalities related to a depressive episode, including psychotherapy or pharmacotherapy.

Participants will undergo baseline questionnaires before completing four daily smartphone-based assessments over seven consecutive days, evaluating their emotion beliefs, emotion regulation, and emotional outcomes. Participants will be randomly assigned to either the intervention or the monitoring-only control group. Following a four-day break, participants in the intervention group will receive a valence-specific ecological momentary intervention targeting emotion regulation in daily life. During this period, participants will report their emotional experiences twice daily and will be supported in implementing either reappraisal or savoring strategies based on the valence of their current predominant emotion. Participants in the control group will be instructed to complete two daily assessments, monitoring their emotions and the strategies used to regulate them. After an additional four-day break, participants will be invited to complete post-assessment questionnaires capturing emotion regulation ability, self-efficacy and strategy use, depressive symptoms, emotion beliefs (controllability, usefulness), and another week of ecological momentary assessment (four per day), encompassing, among other variables, the use of emotion regulation strategies and the experience of positive and negative emotions.

Hypotheses:

The valence-specific intervention is hypothesized to enhance emotion regulation ability and self-efficacy, emotional outcomes (depressive symptoms, positive and negative affect), and emotion beliefs (controllability, usefulness) and to increase the application of reappraisal in negative and savoring in positive emotional contexts in daily life.

The investigators hypothesize that individuals with current depressive disorders will report more unfavorable beliefs about emotions and higher use of strategies associated with dampening positive emotions compared to controls at baseline.

Furthermore, the investigators expect that unfavorable beliefs about positive emotions at baseline (i.e., assuming that positive emotions are harmful) may predict the selection of dampening strategies in the context of positive emotions.

ELIGIBILITY:
Inclusion Criteria:

* Online consent for participation
* Adequate proficiency in the German language, encompassing both reading and comprehension skills
* Ownership of a smartphone, compatible with either Android or iOS operating systems, and access to the Internet

For individuals in the clinical group with current depressive disorders:

* Currently meeting the DSM-5 criteria for a mild or moderate major depressive episode, or persistent depressive disorder

Exclusion Criteria:

* Current severe substance use disorder
* Acute suicidality
* Current severe major depressive episode
* Lifetime bipolar disorder
* Lifetime psychotic disorders

For the control group, additional exclusion criteria include:

* Meeting the DSM-5 criteria for a major depressive episode within the last 12 months
* History of severe major depressive episodes
* Recurrent depressive disorder
* History of persistent depressive disorder
* Current treatment (psychotherapy, pharmacotherapy) for depressive symptoms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Emotion Regulation Ability (Positive, Negative Emotions) | 0 weeks, 3 weeks
  The Perth Emotion Regulation Competency Inventory (PERCI; Preece al., 2021) consists of 32 items, rated on a 7-point scale (1 = strongly disagree, 4 = neither agree nor disagree, 7 = strongly agree) and measures people's ability to regulate their positive and negative emotions. Two different composite scores can be computed to indicate positive and negative emotion regulation ability (Min = 16, Max = 112 for each score), with higher scores indicating a higher level of difficulty regulating positive or negative emotions.
Emotion Regulation Self-Efficacy for Positive and Negative Emotions | 0 weeks, 3 weeks
  The German version of the Regulatory Emotional Self-Efficacy-Revised (RESE-R) Scale (adapted from Caprara et al., 2008) consists of 10 items, rated on a 5-point scale (1 = not at all well to 5 = very well). The scale assesses self-efficacy in expressing positive emotions (4 items, Min = 1, Max = 5) and in managing negative emotions (despondency/distress: 3 Items, anger/irritation: 3 items, Min = 1, Max = 5), with higher scores indicating higher self-efficacy beliefs.

SECONDARY OUTCOMES:
Emotion Regulation Strategy Use in Positive and Negative Emotional Contexts | 0 weeks, 3 weeks
  Data will be collected using an adaption of the smartphone app EmoTrack (adapted from Pruessner et al., 2023). The app assesses among other factors, the intensity with which participants employ various emotion regulation strategies to manage specific positive and negative emotions, using an 11-point scale (1 = not at all, 11 = very much). Scores for strategy usage will be aggregated across all intensity ratings from the four daily measurements over a continuous seven-day period (Min = 1, Max = 11). Higher scores indicate that a participant engages in a specific strategy more strongly in daily life.
Depressive Symptoms | 0 weeks, 3 weeks
  The Beck Depression Inventory-II (Wang et al., 2013) consists of 21 items, rated on a 4-point scale (0-3) with four statements of increasing severity related to a specific depressive symptom. Higher sum scores (Min = 0, Max = 63) indicate a higher severity of depressive symptoms.
Positive and Negative Affect | 0 weeks, 3 weeks
  Data will be collected using an adaption of the smartphone app EmoTrack (adapted from Pruessner et al., 2023). The app measures among other factors, the intensity of specific positive and negative emotions selected from the Positive and Negative Affect Schedule - Expanded Form (PANAS-X; Watson & Clark, 1994), using an 11-point scale (1 = not at all, 11 = very much). Scores for positive and negative emotions will be aggregated across all intensity ratings from the four daily measurements over a continuous seven-day period (Min = 1, Max = 11). Higher scores indicate that participants experience a higher level of positive (resp. negative) emotions in daily life.
Emotion Beliefs (Controllability, Usefulness) about Positive and Negative Emotions | 0 weeks, 3 weeks
  The Emotion Beliefs Questionnaire (EBQ, Becerra et al., 2020) consists of 16 items, rated on a 7-point scale (1 = strongly disagree, 4 = neither agree nor disagree, 7 = strongly agree). Sum scores can be computed for different subscales: General-Contollability (8 Items, Min: 8; Max: 56), Positive-Usefulness (4 Items, Min: 4, Max: 28), Negative-Usefulness (4 Items, Min: 4, Max: 28), with higher scores indicating that people believe, that emotions are uncontrollable and useless.

OTHER OUTCOMES:
Well-being | 0 weeks, 3 weeks
  The World Health Organization Well-Being Index (WHO-5; Topp et al., 2015) consists of 5 items, rated on a 6-point scale (0 = at no time, 5 = all of the time). Elevated scores indicate a higher well-being (Min = 0, Max = 25).
Life Satisfaction | 0 weeks, 3 weeks
  The Satisfaction With Life Scale (SWLS; Diener et al., 1985) comprises 5 items, rated on a 7-point scale (1 = strongly disagree to 7 = strongly agree). Higher scores indicate a higher level of life satisfaction (Min = 5, Max = 35).
Emotion Beliefs about Positive Emotions (Delay Happiness, Living in the Moment) | 0 weeks, 3 weeks
  The Delaying Happiness and Living in the Moment Scale (Park et al., 2021) consists of 2 subscales with 10 items each, rated on a 7-point scale (1 = strongly disagree to 7 = strongly agree). Higher values indicate stronger beliefs that happiness is an investment over time (Delay Happiness) or stronger beliefs that one should savor happiness now versus later (Living in the Moment, Min = 1, Max = 7 for each scale).
Emotion Beliefs about Positive Emotions (Fear of Happiness) | 0 weeks, 3 weeks
  The Fear of Happiness Scale (Joshanloo et al., 2014) consists of 5 items. Each item is measured on a 7-point scale (1 = strongly disagree to 7 = strongly agree). Higher scores indicate a greater fear of happiness (Min = 5, Max = 35).
Negative Emotional Contrast Avoidance | 0 weeks, 3 weeks
  The Contrast Avoidance Questionnaire-General (CAQ-GE; Llera et al., 2017) consists of 25 items, answered on a 5-point scale (1 = not at all true, 2 = slightly true, 3 = somewhat true, 4 = very true, and 5 = absolutely true), which are assigned to two subscales. Higher scores on the two subscales indicate a higher tendency to create and sustain negative emotions to avoid negative emotional contrasts (18 items, Min = 18, Max = 90) and more discomfort with emotional shifts (7 items, Min = 7, Max = 35).
Emotion Regulation Strategy Use | 0 weeks, 3 weeks
  The Heidelberg Form for Emotion Regulation Strategies (HFERST; Izadpanah et al., 2019) consists of 28 items that measure the habitual use of a range of emotion regulation strategies on a 5-point scale (1 = never, 2 = occasionally, 3 = about half the time, 4 = usually, 5 = always): rumination, avoidance, expressive suppression, experience suppression, reappraisal, social support, acceptance, and problem solving. Higher responses indicate a more frequent use of the specific emotion regulation strategy (Min = 1, Max = 5 for each scale).
Self-Esteem | 0 weeks, 3 weeks
  The Rosenberg Self-Esteem Scale (RSES; Roth et al., 2008) consists of 10 items, rated on a 6-point Likert scale (1 = strongly disagree to 6 = strongly agree). Higher score indicate a higher level of self-esteem (Min = 1, Max = 6).
Locus of Control | 0 weeks, 3 weeks
  The Internal-External Locus of Control-4 (IE-4; Niessen et al, 2022) Scale comprises 4 items, rated on a 5-point scale (1 = doesn't apply at all, 2 = applies a bit, 3 =applies somewhat, 4 = applies mostly, 5 = applies completely). The items can be allocated to two subscales: Internal Locus of Control (IL) and External Locus of Control (EL). Elevated scores on the Internal Locus of Control subscale signify a stronger belief in personal control over life events, whereas higher scores on the External Locus of Control subscale indicate a perception that events occur due to chance, fate, or the influence of powerful others
Controllability Beliefs about Emotions | 0 weeks, 3 weeks
  The Implicit Theories of Emotion Scale (Tamir et al., 2007) consists of 5 items, answered on a 5-point scale (1 = strongly disagree, 5 = strongly agree). Higher scores indicate that a person believes emotions are malleable and controllable (Min = 1, Max = 5).
Anxiety Symptoms | 0 weeks, 3 weeks
  The General Anxiety Disorder Scale (GAD-7; Spitzer et al., 2006) consists of 7 items, rated on a 4-point scale (0 = not at all, 1 = several days, 2 = more than half the days, 3 = nearly every day). Scores range from 0 to 21, with higher scores indicating a higher severity of symptoms of generalized anxiety disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Ilka Mueller, M.Sc., Principal Investigator — Department of Psychology, Heidelberg University; Luise Pruessner, M.Sc., Principal Investigator — Department of Psychology, Heidelberg University; Steffen Hartmann, M.Sc., Principal Investigator — Department of Psychology, Heidelberg University; Sven Barnow, PhD, Study Chair — Department of Psychology, Heidelberg University
Locations (1):
- Department of Clinical Psychology and Psychotherapy, Institute of Psychology, Heidelberg University, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
De-identified dataset
Supporting Information: SAP, Analytic Code
Time Frame: Data will be made available after the publication of the study results.
Access Criteria: Open access, available upon request.
URL: https://osf.io/

REFERENCES:
- [Background] Park LE, Fujita K, Naragon-Gainey K, Radsvick TM, Jung HY, Xia J, Ward DE, Paravati E, Weng J, Italiano A, Valvo A. Happiness-To enjoy now or later? Consequences of delaying happiness and living in the moment beliefs. Emotion. 2023 Feb;23(1):138-162. doi: 10.1037/emo0000850. Epub 2021 Nov 15. PMID 34780240
- [Background] Izadpanah S, Barnow S, Neubauer AB, Holl J. Development and Validation of the Heidelberg Form for Emotion Regulation Strategies (HFERST): Factor Structure, Reliability, and Validity. Assessment. 2019 Jul;26(5):880-906. doi: 10.1177/1073191117720283. Epub 2017 Jul 21. PMID 28730850
- [Background] Llera SJ, Newman MG. Development and validation of two measures of emotional contrast avoidance: The contrast avoidance questionnaires. J Anxiety Disord. 2017 Jun;49:114-127. doi: 10.1016/j.janxdis.2017.04.008. Epub 2017 Apr 28. PMID 28500921
- [Background] Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. Psychother Psychosom. 2015;84(3):167-76. doi: 10.1159/000376585. Epub 2015 Mar 28. PMID 25831962
- [Background] Roth M, Altmann T. A Comparison of the Predictive Validity of Self-Esteem Level and Directly Measured Self-Esteem Stability in the Temporal Prediction of Psychological Distress. Front Psychol. 2020 Jul 24;11:1770. doi: 10.3389/fpsyg.2020.01770. eCollection 2020. PMID 32849049
- [Background] Becerra R, Preece DA, Gross JJ. Assessing beliefs about emotions: Development and validation of the Emotion Beliefs Questionnaire. PLoS One. 2020 Apr 14;15(4):e0231395. doi: 10.1371/journal.pone.0231395. eCollection 2020. PMID 32287328
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Background] Joshanloo M, Lepshokova ZK, Panyusheva T, Natalia A, Poon WC, Yeung, VWL, ... & Jiang DY. Cross-cultural validation of Fear of Happiness Scale across 14 national groups. Journal of Cross-Cultural Psychology. 2014; 45(2): 246-264.
- [Background] Preece DA, Becerra R, Sauer-Zavala S, Boyes M, McEvoy P, Villanueva C, Ibonie S, Gruber J, Hasking P, Gross JJ. Assessing Emotion Regulation Ability for Negative and Positive Emotions: Psychometrics of the Perth Emotion Regulation Competency Inventory in United States Adults. J Affect Disord. 2021 Nov 1;294:558-567. doi: 10.1016/j.jad.2021.07.055. Epub 2021 Jul 16. PMID 34330052
- [Background] Caprara GV, Di Giunta L, Eisenberg N, Gerbino M, Pastorelli C, Tramontano C. Assessing regulatory emotional self-efficacy in three countries. Psychol Assess. 2008 Sep;20(3):227-37. doi: 10.1037/1040-3590.20.3.227. PMID 18778159
- [Background] Watson D, Clark LA. The PANAS-X: Manual for the Positive and Negative Affect Schedule - Expanded Form [Unpublished Manuscript] University of Iowa. 1994.
- [Background] Wang YP, Gorenstein C. Psychometric properties of the Beck Depression Inventory-II: a comprehensive review. Braz J Psychiatry. 2013 Oct-Dec;35(4):416-31. doi: 10.1590/1516-4446-2012-1048. Epub 2013 Dec 23. PMID 24402217
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Niessen D, Schmidt I, Groskurth K, Rammstedt B, Lechner CM. The Internal-External Locus of Control Short Scale-4 (IE-4): A comprehensive validation of the English-language adaptation. PLoS One. 2022 Jul 11;17(7):e0271289. doi: 10.1371/journal.pone.0271289. eCollection 2022. PMID 35816496